CLINICAL TRIAL: NCT06619015
Title: The Impact of Pramlintide on Top of Semaglutide in Obese People With Prediabetes
Brief Title: Tailoring Obesity Treatment Trial
Acronym: TOTT
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Awaiting approval from the Danish medical agency
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24/39715; 2024-510802-10-00 (EU CTIS Number)
Record Dates: First submitted 2024-08-28; First posted 2024-10-01 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: Obesity; Appetite Regulation; PreDiabetes
Keywords: semaglutide; pramlintide; symlin; placebo; obesity; individualized medicine; tailoring treatment; Anti-Obesity Drugs; Appetite Regulation; Treatment Effect Heterogeneity; PreDiabetes
MeSH Terms: conditions — Obesity; Prediabetic State | interventions — pramlintide; semaglutide; Sodium Chloride

STUDY DESIGN:
Intervention Model Description: All subjects will receive weekly semaglutide inj. for 26 weeks. After 24 weeks of treatment, the subjects will be randomized to receive either pramlintide or placebo, in addition to semaglutide for the last two weeks of the study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Semaglutide and placebo (Active Comparator): All subjects will receive weekly semaglutide inj. for 26 weeks. After 24 weeks of treatment, this group will be randomized to receive placebo, in addition to semaglutide for the last two weeks of the study.
  Interventions: Drug: Semaglutide Pen Injector; Drug: Sodium Chloride 0.9% Inj
- Semaglutide and pramlintide (Experimental): All subjects will receive weekly semaglutide inj. for 26 weeks. After 24 weeks of treatment, this group will be randomized to receive pramlintide, in addition to semaglutide for the last two weeks of the study.
  Interventions: Drug: Pramlintide Acetate 1 MG/ML; Drug: Semaglutide Pen Injector

INTERVENTIONS:
Drug: Pramlintide Acetate 1 MG/ML — Symlin (R) (Pramlintide acetate) 1000mcg/ml, will be administered as a continuous infusion at a rate of 15mcg/hour, equivalent to the daily recommended maximum dosage of 360mcg/day.
  Other Names: Symlin
  Arms: Semaglutide and pramlintide
Drug: Semaglutide Pen Injector — Semaglutide from 0,25mg/week to 2,4mg/week
  Other Names: Wegovy
Drug: Sodium Chloride 0.9% Inj — Placebo
  Other Names: isotonic saline solution
  Arms: Semaglutide and placebo

SUMMARY:
The two main aims of this clinical study is;

1. To investigate if the results from a series of physiological tests and questionnaires prior to treatment, can be used to predict the treatment response to obesity medication
2. To investigate the effect of combining semaglutide and pramlintide on various aspects of appetite, food preference and eating habits.

The study is planed as a 26 week, double blinded, randomized, placebo controlled trial. The goal is to include N=40. They will all receive weekly semaglutide injections. After 24 weeks they will be randomized to receive either an amylin analog (pramlintide) or placebo as a continuous infusion for two weeks, in addition to weekly semaglutide.

The results from this study will contribute to identifying possible predictors of treatment response, enabling optimal individualized medical weight loss treatment. As well as providing knowledge on the complex interplay between incretin hormones and their effects on appetite and eating habits.

DETAILED DESCRIPTION:
Obesity is a major global health challenge and the prevalence of obesity is increasing. Presence of obesity increases the risk of several diseases, physical limitations and an increased mortality. When weightloss is wanted in order to avoid or treat some of these diseases, medical weight loss treatment is one of the options. Among these modified gut hormones, such as Glucagon Like Peptide -1 Receptor agonists (GLP-1RA). However, the individual response to GLP-1RA treatments varies considerably. Currently the best predictor of total weight loss is achieved weight loss after three months of treatment. With more pharmaceutical options to come, a trial and error approach is not appropriate. There is a need to identify possible pre-treatment predictors to treatment response.

This is one of the project's main aims. By being able to predict the treatment response, one can tailor the obesity treatment to the individual improving the treatment outcome.

Amylin is co-secreted with insulin from the pancreas in response to meals. It is found to have many similar effects in the body as GLP-1. However their combination, especially on appetite, food preferences and eating pattern is sparsely investigated. This is the other main aim of the project.

This clinical study will be a 26 week, randomized, double-blinded, placebo-controlled trial. Forty overweight (BMI ≥30kg/m2) individuals with pre-diabetes (HbA1c 39-47 mmol/mol) will all receive once-weekly semaglutide for 26 weeks. Semaglutide will be given in escalating doses aiming to reach the maximal dose of 2.4 mg (maximum dosage approved for treatment of overweight), but accepting lower maximal tolerable dosage.

After 24 weeks of treatment, they will be stratified according to their weight loss (<15% or ≧15%) and based on this stratification, block randomized 1:1 to receive either pramlintide or placebo(normal isotonic 0.9% saline solution) in addition to weekly semaglutide. Pramlintide will be continuously infused, starting at a dosage of 7,5 mcg/hour for three days, and if tolerated, the dosage will be increased to 15 mcg/hour for the remaining eleven days. Previous studies have found measurable changes in appetite after a single dosage of pramlintide, and measurable weight loss after two weeks of treatment. For the continuous infusion a commercially available insulin pump will be used.

At study start and, prior to semaglutide treatment, body composition, REE and gastric emptying rate will be measured. Various aspects of appetite will be assessed by the results from the meal tests, the "taste test", appetite assessment and eating related questionnaires. An appetite Visual Analog Scale (VAS) will be measured prior to, and following the standardized meal test and the ad libitum meal test. Satiety will be assessed by a VAS following the standardized meal test. Appetite related sensory specific desire will be assessed by the participants rating of a "taste test" consisting of a variety of small food samples representing the sensory profiles of sweet, sour, salt, bitter, fat, umami/savory and spicy, respectively. The "taste test" will be performed prior to the ad libitum test and as previously described. And satiation will be assessed by measuring calories consumed to reach fullness and terminate the meal at the ad libitum meal test. While the Food pleasure scale, Yale Food Addiction Scale 2.0, Dutch Eating Behavior Questionnaire and The Eating Disorder Quality of Life Scale questionnaires will assess hedonic, emotional and binge- eating patterns and eating related quality of life. The combined results of these physical measurements, questionnaires, appetite and hunger assessments will be used to identify the participants' main obesity driver or obesity "phenotype" similarly as previously described.

These tests will be repeated at the end of the study and the results compared. The "taste test" and ad libitum meal test will also be performed after 24 weeks, prior to the addition of either pramlintide or placebo.

Additionally blood samples will be taken at baseline, after 24 weeks and at the end of the study, measuring biomarkers related to metabolism, bone metabolism and organ specific biomarkers.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≧ 30kg/m2
* HbA1c 39-47 mmol/mol (pre-diabetes)
* Male or female
* Aged >18 years of age and <70 years
* Negative pregnancy test, and willing to use contraceptives during the study period

Exclusion Criteria:

* Presence of diabetes with or without treatment
* Current or recent (<6 months) treatment with GLP1 RA's
* Previous gastrointestinal surgery that might affect gastric emptying, nutritional absorption and postprandial GI peptide production
* History of acute or chronic pancreatitis
* Chronic kidney disease
* Use of any antipsychotic drugs
* Use of any antiresorptive or bone-anabolic drugs or fractures within < 6 months
* Use of systemic oral glucocorticoids within < 6 months
* Newly (< 3 months) initiated hormonal contraceptive or other hormone therapy
* Recent (<3 months) weight loss ≧ 1% of body weight
* Presence of Binge eating disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change in kilocalorie (kCal) consumption at ad libitum meal test, from baseline, to after 26 weeks of semaglutide of which the last two weeks is with the addition of either pramlintide or placebo | From baseline at the start of the study(week 0), to the end of the study after 26 weeks

SECONDARY OUTCOMES:
Difference in total weight loss between the subgroups (Obesity phenotypes) | From baseline (week 0) to end of study (week 26)
Change in appetite and satiety sensations as measured by Visual Analog Scale (VAS) prior to and following the meal tests | From baseline(week 0) to after 24 weeks, and to the end of the study(week 26)
  The meal test will be performed at baseline, after 24 weeks and at the end of the study(week 26). Prior to and following the meal tests a VAS measuring appetite and satiety sensation will be answered.
Change in gastric emptying rate assessed by paracetamol (acetaminophen) test | From baseline (week 0) to end of study(week 26)
  The gastric emptying test will be performed at baseline (week 0) and at the end of the study (week26).
Total weight loss | From baseline(week 0) to after 24 weeks, and to the end of the study(week 26)
  Total weight loss from baseline, after 24 weeks, and at the end of the study( week 26) The results will be repoted as percentage (%) weight loss.
Total weight loss | From baseline(week 0) to after 24 weeks, and to the end of the study(week 26)
  Total weight loss from baseline, after 24 weeks, and at the end of the study( week 26) The results will be repoted as total weight loss in Kg

OTHER OUTCOMES:
Change in sensory specific desires as measured by a taste test | From baseline (week 0) to after 24 weeks, and to the end of the study (week 26)
  The taste test will be performed at baseline, after 24 weeks, and at the end of the study (week 26)
Change in hedonic eating behavior as measured by questionnaires | From baseline (week 0) to after 24 weeks, and to the end of the study (week 26)
  The questionnaires; Food pleasure scale, Yale Food Addiction Scale 2.0, Dutch Eating Behavior Questionnaire and The Eating Disorder Quality of Life Scale questionnaires will assess hedonic, emotional and binge- eating patterns and eating related quality of life. The questionnaires will be answered at baseline(weeks 0) , after 24 weeks and at the end of the study (week 26)

CONTACTS AND LOCATIONS:
Overall Officials: Claus Bogh Juhl, MD, phd, professor, Principal Investigator — Head of endocrinology dept.
Locations (1):
- University hospital of Southern Denmark, Esbjerg, Denmark